CLINICAL TRIAL: NCT07003035
Title: A Multi-Center Prospective Cohort Study on the Clinical Advantages of Personalized Total Knee Arthroplasty System
Brief Title: A Multi-Center Study on the Clinical Advantages of Personalized Total Knee Arthroplasty System
Status: Not yet recruiting | Type: Observational
Sponsor: YujiakuoTHU (Other)
Collaborators: Peking University Shougang Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor-Investigator, YujiakuoTHU, Prof., Beijing Tsinghua Chang Gung Hospital
Organization: Beijing Tsinghua Chang Gung Hospital (Other)
Other Study IDs: 23705-4-02
Record Dates: First submitted 2025-03-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: A total of 80 participants will be enrolled, with 40 receiving personalized total knee arthroplasty and 40 receiving conventional TKA. Participants will be followed for one year post-surgery to assess clinical outcomes.

SUMMARY:
The purpose of this study is to evaluate the clinical benefits of personalized total knee arthroplasty (TKA) in comparison with conventional TKA. The study aims to assess surgical outcomes, functional recovery, complication rates, and cost-effectiveness in a multi-center, prospective cohort study.

DETAILED DESCRIPTION:
This study builds on long-term research on the design, manufacturing, and validation of personalized total knee arthroplasty (TKA) prostheses . The clinical study aims to assess the performance of the femoral, tibial, and meniscal components within a personalized TKA system.

This is a prospective cohort and controlled study involving 80 patients, including 40 in the experimental group and 40 in the control group. Participants will be 50-80 years old, diagnosed with end-stage knee osteoarthritis, post-traumatic arthritis, avascular necrosis, inflammatory arthritis, or deformities requiring total knee arthroplasty. They will be followed for one year post-surgery to assess clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50-80 years.
2. Diagnosed with end-stage knee osteoarthritis, post-traumatic arthritis, avascular necrosis, or inflammatory arthritis requiring total knee arthroplasty.
3. Willing and able to provide informed consent.

Exclusion Criteria:

1. History of prior knee surgery or knee replacement.
2. Severe knee deformity (valgus >20° or varus >15°) or instability.
3. Severe contracture (>25° flexion contracture).
4. Undergoing total knee revision surgery.
5. Rheumatoid arthritis diagnosis.
6. BMI >35.
7. Neuromuscular disorders affecting knee stability or gait.
8. Pregnancy or lactation.
9. Presence of significant comorbidities posing unacceptable risk, including but not limited to metabolic, renal, hepatic, pulmonary, cardiac, hematologic, neurological, endocrine, infectious, or gastrointestinal conditions.
10. Active or recent severe infections or malignancy.
11. History of drug or alcohol abuse in the past six months.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will recruit adult patients aged 50-80 years who are undergoing total knee arthroplasty for end-stage knee osteoarthritis or related conditions. Participants will be selected from multiple hospital centers to ensure a diverse patient population.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | At baseline, 6 months, and 12 months post-surgery
  The Knee Society Score is a standardized assessment tool to evaluate pain, range of motion, and functional ability following total knee arthroplasty. It includes two sub-scores: a clinical knee score and a functional score.
  Each sub-score ranges from 0 to 100, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Pain Severity - Visual Analog Scale (VAS) | At baseline, 6 months, and 12 months post-surgery.
  Pain severity will be measured using the VAS, a 10 cm horizontal line ranging from 0 (no pain) to 10 (worst imaginable pain).
  Higher scores indicate worse pain.
Pain Severity - Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | At baseline, 6 months, and 12 months post-surgery
  Pain will also be assessed using the WOMAC Pain Subscale, part of the validated WOMAC Index for knee osteoarthritis.
  Each item is scored from 0 to 4, and the subscale total ranges from 0 (no pain) to 20 (maximum pain).
  Higher scores indicate worse pain.
Functional Improvement - SF-36 Health Survey | At baseline, 6 months, and 12 months post-surgery.
  Physical function will be assessed using the 36-Item Short Form Health Survey (SF-36). The Physical Functioning domain is scored from 0 to 100, with higher scores indicating better health-related quality of life.
Functional Improvement - Knee Injury and Osteoarthritis Outcome Score (KOOS) | At baseline, 6 months, and 12 months post-surgery
  The KOOS is a validated tool assessing knee function across five domains. Each domain score ranges from 0 to 100, with higher scores indicating better knee function and fewer symptoms.
Functional Improvement - Gait Analysis | At baseline, 6 months, and 12 months post-surgery
  Gait performance will be evaluated using temporospatial parameters such as gait speed (m/s), step length (cm), and cadence (steps/min), measured using standardized motion capture or pressure-sensitive walkways.
Prosthesis Positioning and Alignment | At baseline and 12 months post-surgery.
  Radiographic evaluation will assess implant positioning and limb alignment.
Surgical Complication Rate | At 12 months post-surgery.
  The rate of postoperative complications including infections, deep vein thrombosis (DVT), and revision surgeries will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China